CLINICAL TRIAL: NCT02905539
Title: A Randomized, Double-blind Comparative Study Comparing Ferric Carboxymaltose (Ferinject) and Iron Isomaltoside 1000 (Monofer) for Iron Substitution in Iron-deficiency Anemia
Brief Title: A Study Comparing the Iron Substitution With the Medicinal Products Ferinject or Monofer
Acronym: HOMe_aFers_1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-0101; 2015-004808-36 (EudraCT Number); U1111-1176-4563 (Registry Identifier: WHO Universal Trial Number); DRKS00010766 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2019-04

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Iron; anemia; phosphorus; FGF-23
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — iron isomaltoside 1000; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron Isomaltoside 1000 (Experimental): Subjects receive Iron Isomaltoside 1000 solution intravenously. Dosage: A unique dose of 20 mg per kilogram bodyweight, but total dose is not more than 1000 mg.
  Interventions: Drug: Iron Isomaltoside 1000
- Ferric Carboxymaltose (Active Comparator): Subjects receive Ferric Carboxymaltose solution intravenously. Dosage: A unique dose of 20 mg per kilogram bodyweight, but total dose is not more than 1000 mg.
  Interventions: Drug: Ferric Carboxymaltose

INTERVENTIONS:
Drug: Iron Isomaltoside 1000
  Other Names: Monofer
  Arms: Iron Isomaltoside 1000
Drug: Ferric Carboxymaltose
  Other Names: Ferinject
  Arms: Ferric Carboxymaltose

SUMMARY:
The purpose of this study is to determine to what extend a treatment with the iron compounds Iron Isomaltoside 1000 or Ferric Carboxymaltose is leading to hypophosphatemia and to study the potential clinical impact of hypophosphatemia.

DETAILED DESCRIPTION:
Recent studies suggested that intravenous iron preparations for anemia treatment may have adverse effects on phosphorus regulation, as they may induce an increase in the phosphaturic hormone Fibroblast Growth Factor-23 (FGF-23) and a subsequent fall in plasma phosphorus levels.

So far it is unknown if these effects are class- or substance-specific.

This study will address the question whether among female participants with iron deficiency anemia the application of ferric-(III)-derisomaltose and ferric carboxymaltose will cause episodes of hypophosphatemia to same extend. The investigators will additionally compare the effects of the two iron preparations on other parameters of calcium-phosphate metabolism, and decipher potential consequences of hypophosphatemia by analysing cardiac function, immunological parameters and quality of life.

In order to investigate these outcomes, 60 women with iron deficient anemia will be randomised to receive either ferric-(III)-derisomaltose or ferric carboxymaltose.

The monocentric study will be conducted at Saarland University Medical Center. For each participating woman, the study comprises five visits to the study center during a period of five weeks.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent,
* female,
* gynecological blood losses,
* age ≥ 18 years,
* iron deficiency anemia,
* Hemoglobin < 12,0 g/dl,
* Serum-Ferritin ≤ 100 ng/ml or Serum-Ferritin ≤ 300 ng/ml and Transferrin-saturation ≤ 30 %,
* Intolerance to or inefficacy of an oral iron supplement
* estimated Glomerular Filtration Rate > 15 ml/min/1.73 m²

Exclusion Criteria:

* known hypersensitivity to MonoFer® or FERINJECT®,
* severe, known hypersensitivity to other intravenous iron preparations,
* Plasma Phosphate < 2.5 mg/dl at screening,
* Hemochromatosis,
* Untreated hyperparathyroidism,
* Renal replacement therapy/kidney transplantation,
* Active malignant disease, disease-free survival for less than 5 years,
* Intravenous iron administration within the last 30 days,
* Treatment with erythropoietin or erythropoietin-stimulating agents, transfusion of red blood cells, radiotherapy or chemotherapy within the last 60 days,
* Surgery under anesthetic within the last 10 days,
* Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 fold above levels in healthy individuals,
* Acute febrile infections within the last 7 days,
* Chronic inflammatory diseases requiring a systemic antiinflammatory treatment,
* self-reported severe asthma or eczema,
* presence of relative contraindications (any allergy, any immunologic or inflammatory disease, history of atopic allergies), for which a treatment with the medicinal investigational products is not deemed indicated by the investigator,
* pregnancy,
* women of childbearing potential without an effective method of contraception,
* lactating women,
* Present alcohol or drug dependency,
* Patients with a history of a psychological illness or seizures,
* Non-compliance or administration of any investigational drug within 30 days preceding the study start.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Incidence of hypophosphatemia | From baseline to day 35
  The incidence of hypophosphatemia is defined as a drop of serum phosphate below 2.0 mg/dl.

SECONDARY OUTCOMES:
Changes of plasma phosphate concentrations. | From baseline to day 35
Changes of fractional Phosphate urinary excretion. | From baseline to day 35
Changes of Plasma Vitamin D (active, inactive). | From baseline to day 35
Changes of fibroblast growth factor 23 (intact and c-terminal). | From baseline to day 35
Changes of parathyroid Hormone. | From baseline to day 35
Changes of Plasma calcium. | From baseline to day 35
Changes of Plasma alkaline Phosphatase. | From baseline to day 35
Changes of Plasma soluble Klotho. | From baseline to day 35
Changes of Plasma Hepcidin-25. | From baseline to day 35
Changes of Serum N-Terminal Propeptide of Type I Collagen (PINP). | From baseline to day 35
Changes of Pyridinoline (PYD) in the urine | From baseline to day 35
Changes of Quality of life. | From baseline to day 35
  German Version of the Short Form (36) Health Survey by Matthias Morfeld, Inge Kirchberger, Monika Bullinger.
Incidence of (supra)ventricular cardiac arrhythmias in the ambulatory Electrocardiography. | Before and 7 days after administration of iron compound
Changes of QT-time in the 12-lead Electrocardiography. | From baseline to day 35
Changes of QT-Dispersion in the 12-lead Electrocardiography. | From baseline to day 35
Changes of Left Ventricular Mass Index | From baseline to day 7
  Echocardiographic measurement
Count of monocyte subpopulations. | Right before the singular infusion of the iron compound is started and right after infusion of the iron compound is completed.
  Count of classical , intermediate and nonclassical monocytes using flow cytometry.
Measurement of phagocytic capacity of monocytes. | Right before the singular infusion of the iron compound is started and right after the infusion of iron compound is completed.
  Exposition of Monocytes to Fluoresbrite Yellow Green (YG) Carboxylate Microspheres and subsequent flow cytometric count of Fluorescein isothiocyanate-positive Monocytes.
Changes of fatigue | From baseline to day 35
  The German Version of the Multidimensional Fatigue Inventory. (Smets E. M. A., Garssen B., Bonke B. and Haes de J. C. J. M. (1995). The Multidimensional Fatigue Inventory (MFI); Psychometric qualities of an instrument to assess fatigue. Journal of Psychosomatic Research, 39, 315-325.)
Changes of Left Atrial Volume Index | From Baseline to day 7
  Echocardiographic measurement
Changes of Systolic Ejection Fraction | From Baseline to day 7
  Echocardiographic measurement
Changes of Diastolic Left Ventricular Function | From Baseline to day 7
  Echocardiographic measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Heine, MD, Principal Investigator — Universität des Saarlandes; Danilo Fliser, MD, Study Director — Universität des Saarlandes
Locations (1):
- Universitätsklinikum des Saarlandes, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emrich IE, Lizzi F, Siegel JD, Seiler-Mussler S, Ukena C, Kaddu-Mulindwa D, D'Amelio R, Wagenpfeil S, Brandenburg VM, Bohm M, Fliser D, Heine GH. Hypophosphatemia after high-dose iron repletion with ferric carboxymaltose and ferric derisomaltose-the randomized controlled HOMe aFers study. BMC Med. 2020 Jul 13;18(1):178. doi: 10.1186/s12916-020-01643-5. PMID 32654663